CLINICAL TRIAL: NCT04306497
Title: Clinical Trial of TCM Differentiation and Treatment Protocol of COVID-19 in Jiangsu Province
Brief Title: TCM Differentiation and Treatment Protocol of COVID-19
Acronym: TDATPOC
Status: Completed | Type: Observational
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JSZYJ202001
Record Dates: First submitted 2020-03-01; First posted 2020-03-13 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: COVID-19; Syndrome investigation; differentiation treatment; multicenter cohort study
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort of western medicine: 1. Routine treatment：
     ① support treatment:maintain water and electrolyte balance .
     ②oxygen therapy: give nasal catheters to inhale oxygen.
     ③ basic treatment of traditional Chinese and western medicine: antiviral drugs and proprietary Chinese medicines with similar composition or function to the observed scheme of differentiation and treatment of traditional Chinese medicine are not included in the scope of such drugs.
  2. Antiviral drugs ：Clinicians can judge according to the patient's condition according to the latest version of the diagnosis and treatment plan for COvID-19 issued by the General Office of the National Health Commission / the Office of the State Administration of traditional Chinese Medicine (currently the latest version is the sixth trial edition). Select any of the recommended antiviral drugs(for example:IFN-α、lopinavir-ritonavir、Ribavirin、Chloroquine Phosphate、Arbidol)or a combination of two antiviral drugs.
  Interventions: Drug: TCM prescriptions
- Cohort of integrated TCM and western medicine: routine treatment + Antiviral drugs + the following TCM regimens. 1.TCM regimens:① Early stage: Dampness trapped in exterior and interior. Recommended prescription: Huoxiang 15g, Suye15g, Cangzhu15g, Houpo10g, Qianhu15g, Chaihu15g, Huangqin10g, Qinghao20g, Xingren10g, JInyinhua15g, Lianqiao15g.
  Take decocted or granule, one dose a day.
  ② Middle stage: Dampness-toxicity blocking lung Recommended prescription: Zhimahuang9g, Xingren10g, Sangbaipi30g, Tinglizi20g, Dongguazi20g, Fabanxia10g, Houpo10g, Suzi15g, Baijiezi10g, Gualoupi15g, Xuanfuhua9g, Xiangfu10g, Yujin10g, Taoren10g, Huangqi20g.
  Take decocted or granule, one dose a day.
  Interventions: Drug: TCM prescriptions

INTERVENTIONS:
Drug: TCM prescriptions — TCM prescriptions1:Take decocted or granule, one dose a day; TCM prescriptions2:Take decocted or granule, one dose a day.

SUMMARY:
Evaluation of the efficacy and safety of TCM differential treatment of COVID-19 in Jiangsu Province based on the historical prospective multicenter cohort study.

DETAILED DESCRIPTION:
This is a multi-center cross-sectional syndrome investigation study, taking confirmed cases as the main observation object, A prospective multicenter cohort study was designed, focusing on the common type with the largest number of confirmed cases, to evaluate the intervention effect of this project in relieving the disEvaluation of the efficacy and safety of TCM differential treatment of COVID-19 inease and preventing disease progressio.

According to the actual situation of receiving treatment, if the subjects received the combination of western medicine and traditional Chinese medicine, it was the exposure group (integrated traditional Chinese and western medicine cohort), and if the subjects only received western medicine treatment, it was the control group (western medicine cohort). The choice of treatment for patients is entirely determined by clinicians according to the patient's condition, and patients are free to choose after fully understanding different schemes).The choice of control group: COVID-19 (common type) who received routine treatment + antiviral therapy；The choice of exposure group: COVID-19 (common type) who received routine treatment + TCM.The sample size is tentatively set at 340.

ELIGIBILITY:
Inclusion Criteria:

* It conforms to the diagnostic criteria of confirmed cases of COVID-19 that belongs to the common type;
* The age ranges from 18 to 80 years old, regardless gender；
* In the prospective study, the patient informed consent and sign the informed consent form (if the subject has no capacity, limited capacity and limited expression of personal will, he or she should obtain the consent of his guardian and sign the informed consent at the same time), the retrospective study is visa-free informed consent.

Exclusion Criteria:

* Women during pregnancy or lactation;
* Allergic constitution, such as those who have a history of allergy to two or more drugs or food, or who are known to be allergic to drug ingredients observed in this study.
* Severe complications such as multiple organ failure and shock occurred.
* Complicated with severe primary diseases such as heart, brain, liver, kidney and so on.
* Patients have mental illness.
* Patients who participated in or is currently participating in other clinical trials within the first month of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It conforms to the diagnostic criteria of confirmed cases of COVID-19.
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
The relief of main symptoms/ disappearance rate of time | 9day
  comparison of the time of relief / disappearance of three main symptoms of fever, cough and shortness of breath
Chest CT absorption | 9day
  with reference to the "pneumonia chest X-ray absorption Evaluation scale" developed by Renyi Yin et al, the final absorption judgment will be used to evaluate the chest CT absorption of patients with pneumonia, which is divided into four levels according to the degree of absorption: complete absorption, majority absorption, partial absorption and no absorption.

SECONDARY OUTCOMES:
Evaluation standard of comprehensive curative effect | 9day
  With reference to the "Therapeutic effect Standard for diagnosis and Syndrome of Traditional Chinese Medicine" and "guiding principles for Clinical Research of New drugs of traditional Chinese Medicine", the final evaluation was based on clinical remission.
Virus antigen negative conversion rate | 9day
  the detection negative rate of nasopharyngeal swab, conjunctival sac secretion virus nucleic acid.
The number of severe and critical conversion cases | 9day
  the number of severe and critical cases occurred after the start of intervention.
Incidence of complications | 9day
  defined as complications during isolation and hospitalization due to pneumonia infected by novel coronavirus, including bacterial infection, aggravation of underlying diseases, etc
Traditional Chinese Medicine Syndrome Score | 9day
  According to the Traditional Chinese Medicine symptom score scale, the change of symptom score before and after treatment was observed.The highest score was 92 points, and the lowest was 23 points. The higher the score, the more severe the symptoms.

OTHER OUTCOMES:
CRP changes | 9day
  Changes in c-reactive protein.
ESR changes | 9day
  Changes in erythrocyte sedimentation rate.
PCTchanges | 9day
  Changes in procalcitonin.
The index of T cell subsets changed | 9day
  Changes of CD4+ and CD8+

CONTACTS AND LOCATIONS:
Locations (1):
- Huai'an fourth people's Hospital, Huaian, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
All researchers in this study